CLINICAL TRIAL: NCT05625165
Title: Epidemiology of Pediatric Traumatology
Acronym: ETP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7956
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-11

CONDITIONS: Fractures in Children
Keywords: Fractures in Children; pediatric fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fractures have been shown to account for 10-25% of injuries in children and the consequences of pediatric fractures are significant and result in significant restriction of activity. Despite this, the epidemiology of pediatric fractures remains poorly detailed.

Investigators seek to establish the incidence of pediatric trauma and fractures and determine patient, trauma and injury characteristics.

ELIGIBILITY:
Inclusion criteria:

* Children treated in the pediatric emergency department of the Strasbourg University Hospitals between January 2014 and December 2020 for skeletal trauma.
* Child and Holders of parental authority who have been informed of the use of their child's data for the purposes of this research and who have not expressed any opposition

Exclusion criteria:

* Patient or legal representative who expressed their opposition to participating in the study
* Impossibility of giving informed information to the subject

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children treated in the pediatric emergency department of the Strasbourg University Hospitals between January 2014 and December 2020 for skeletal trauma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence of pediatric trauma and fractures and to determine the characteristics of patients, traumas and lesions | Files analysed retrospectively from January 01, 2014 to December 31, 2012 will be examined
  This study focuses on retrospective analysis of patients' medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Pédiatrique - CHU de Strasbourg - France, Strasbourg, France